CLINICAL TRIAL: NCT04653090
Title: Varus Stem Positioning Does Not Affect Long-term Functional Outcome in Cementless Anatomical Total Hip Arthroplasty.
Brief Title: Varus Stem Positioning of a Cementless Anatomical THA. (VARABG)
Acronym: VARABG
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: 20.0035
Record Dates: First submitted 2020-11-13; First posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-11

CONDITIONS: Osteoarthritis; Arthroplasty Complications
Keywords: Total hip arthroplasty; varus alignment; anatomical stem; survivorship
MeSH Terms: conditions — Osteoarthritis | interventions — X-Rays

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Varus group: Radiographic stem axis was assessed on standard anteroposterior hip radiographs performed at the 3-month follow-up visit. Alignment was evaluated as described by Reina et al., by the angular deviation of the anatomic femoral axis and the stem axis. The 3 degrees minimal-value was considered to be the threshold defining a varus stem.
  Interventions: Diagnostic Test: Xray
- Neutral group: Alignment between anatomic femoral axis ans stem axis was less than 3°.
  Interventions: Diagnostic Test: Xray

INTERVENTIONS:
Diagnostic Test: Xray — Hip AP Xray

SUMMARY:
Varus positioning is the most common femoral malposition in total hip arthroplasty (THA). The aim of this study was to compare the long-term results of an anatomical cementless femoral stem positioned in varus with those in neutral alignment.

DETAILED DESCRIPTION:
Data were prospectively collected and retrospectively reviewed for all patients who received a cementless anatomical femoral stem in THA between 1998 and 2008. After exclusion criteria applied, 127 stems had an varus axis deviated by more than 3 degrees (varus group) and 156 had an alignment between 0 and 2.9° from the femoral axis (neutral group). Survivorship rates, complications, clinical scores, thigh pain, radiological score, cortical hypertrophy and filling rate were analyzed. Mean follow-up was 10 years.

ELIGIBILITY:
Inclusion Criteria:

* All patients received by several senior surgeons, the same standardized posterolateral total hip arthroplasty, and the same rehabilitation protocol.

Exclusion Criteria:

* Etiologies other than osteoarthritis (osteonecrosis, fracture, dysplasia, rheumatoïd arthritis),
* Complex cases with additional procedure,
* Dual-taper modular or cemented stem,
* Incomplete preoperative data or less than one-year postoperative data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators identified all patients who underwent proximal HA-coated anatomic tapered femoral stem primary THAs between October 1998 and July 2008, through our institutional total joint registry. The data were prospectively collected on the Orthowave© database. This included patients who had an uncemented ABG-2 stem (Stryker, Mahwah, NJ). The study was a test-case retrospective analysis and an institutional review board approval was obtained prior to initiation of the study.
Sampling Method: Non-Probability Sample
Enrollment: 283 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2020-11-05 (Actual)

PRIMARY OUTCOMES:
Long-term survival of THA with varus or neutral cementless fixation of a proximal HA-coated anatomic tapered femoral stem. | Survival evaluation was carried out through study completion at an average of 10 years by the surgeon.
  Kaplan-Meier survivorships free of revision of the femoral component for any reason, femoral fracture and revision of femoral component for fracture were calculated and compared by log-rank test for both group.

SECONDARY OUTCOMES:
Long-term clinical outcomes with varus or neutral femoral stem. | Clinical evaluation was carried out through study completion at an average of 10 years by the surgeon.
  Clinical status was assessed by the Harris hip score (HHS).
Long-term radiological outcomes with varus or neutral femoral stem. | Radiological evaluation was carried out through study completion at an average of 10 years by the surgeon.
  Radiological assessment was conducted at the last follow-up in charge antero-posterior and profile X-Ray.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nîmes, Nîmes, Gard, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reina N, Salib CG, Perry KI, Hanssen AD, Berry DJ, Abdel MP. Mild Coronal Stem Malalignment Does Not Negatively Impact Survivorship or Clinical Results in Uncemented Primary Total Hip Arthroplasties With Dual-Tapered Implants. J Arthroplasty. 2019 Jun;34(6):1127-1131. doi: 10.1016/j.arth.2019.01.055. Epub 2019 Jan 31. PMID 30773361
- [Background] Khalily C, Lester DK. Results of a tapered cementless femoral stem implanted in varus. J Arthroplasty. 2002 Jun;17(4):463-6. doi: 10.1054/arth.2002.32171. PMID 12066277
- [Background] Min BW, Song KS, Bae KC, Cho CH, Kang CH, Kim SY. The effect of stem alignment on results of total hip arthroplasty with a cementless tapered-wedge femoral component. J Arthroplasty. 2008 Apr;23(3):418-23. doi: 10.1016/j.arth.2007.04.002. Epub 2007 Nov 9. PMID 18358382